CLINICAL TRIAL: NCT00304603
Title: A Study to Evaluate the Mode of Action of Topiramate in the Treatment of Obese Subjects With and Without Type 2 Diabetes Mellitus Using DNA Samples From Subjects Who Were Randomized Within Select Previous Topiramate Studies
Brief Title: Mode of Action of Topiramate in the Treatment of Obese Patients With and Without Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003409; TOPMAT-OBE-3001 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC); RWJ-17021-000 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC)
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Obesity; Diabetes Mellitus Type 2
Keywords: Obesity; Type 2 Diabetes Mellitus; Topiramate; Pharmacogenomics; DNA Polymorphism
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients from previous topiramate obesity and diabetes studies: The patients from previous topiramate obesity and diabetes studies (PRI/TOP-INT-31 or PRI/TOP-INT-33 or a subset of patients with diabetes mellitus who were randomized within the PRI/TOP-INT-34 study at sites that also participated in the PRI/TOP-INT-31 study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No treatment was given to the patients as this is an observational study.

SUMMARY:
The purpose of this study is to explore the mode of action of topiramate in the treatment of obese and diabetic patients by testing association between genetic variations within candidate genes or chromosomes (thread like structure found in cell which carries genes) and the clinical outcomes.

DETAILED DESCRIPTION:
This pharmacogenomics (effect of genetic variation on drug response) study will analyze genetic variations in the DNA extracted from blood samples collected from patients who were randomized (assigned to treatments by chance) in 1 of 3 previous topiramate studies on obesity and diabetes. The study consist of a screening telephone contact, a single visit to the study site for a blood sample collection (10 ml of whole blood) for genetic analyses, and a 24-hour post-sample adverse event reporting period. The total duration of the study is 24 hours from the time of the blood sample collection. Safety will be monitored up to 24 hours after blood sample collection. No study medication was administered.

ELIGIBILITY:
Inclusion Criteria:

* Must have been randomized within the previous topiramate obesity and diabetes studies: PRI/TOP-INT-31 or PRI/TOP-INT-33 or a subset of patients with diabetes mellitus who were randomized within the PRI/TOP-INT-34 study at sites that also participated in the PRI/TOP-INT-31 study
* Must consent to participate and use data from previous clinical trials in connection with results from the genetic analyses

Exclusion Criteria:

* Patients who received a blood transfusion within 60 days before collecting DNA samples

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients from previous topiramate obesity and diabetes studies (PRI/TOP-INT-31 or PRI/TOP-INT-33 or a subset of patients with diabetes mellitus who were randomized within the PRI/TOP-INT-34 study at sites that also participated in the PRI/TOP-INT-31 study).
Sampling Method: Probability Sample
Enrollment: 1145 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Percent change in weight | Baseleine to Week 24
  The candidate gene analyses and the genome (entire hereditary information of organism) screen for percent change in weight will be performed in 3 phases. 1) Find polymorphisms (existence of distinctly different types in group of 1 species) within candidate genes and chromosomal regions that impact response to topiramate. 2) Confirm Phase 1 findings. 3) Verify that polymorphisms and chromosomal regions that were associated with percent change in weight in 2 phases are associated with percent change in weight in response to topiramate rather than change in diet and exercise.

SECONDARY OUTCOMES:
Change in in glycosylated hemoglobin (HbA1c) | Baseline to Week 24
Number of patients with central nervous system (CNS) related adverse events | Baseline to Week 24
  Most frequent CNS-related adverse events (ie, paresthesia, depression, difficulty with concentration/attention, anorexia, difficulty with memory, fatigue, somnolence, insomnia, mood problems, and hypoesthesia) and adverse events related to venipuncture are monitored during the study.
Number of patients with adverse events | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study to Explore the Mode of Action of Topiramate in the Treatment of Obese Subjects With and Without Type 2 Diabetes Mellitus Using DNA Samples From Subjects Who Were Randomized Within Select Previous Topiramate Obesity and Diabetes Studies — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=527&filename=CR003409_CSR.pdf